

Title: A Phase 3, Open-label Study to Determine the Long-term Safety and Efficacy of Vedolizumab (MLN0002) in Patients With Ulcerative Colitis and Crohn's Disease

NCT Number: NCT00790933

SAP Approve Date: January 7, 2013

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

# STATISTICAL ANALYSIS PLAN

A Phase 3, Open-label Study to Determine the Long-term Safety and Efficacy of Vedolizumab (MLN0002) in Patients With Ulcerative Colitis and Crohn's Disease

Protocol #: C13008 Amendment 10

SAP Version: Amendment 2 <u>Date of Statistical Analysis Plan:</u> January 7, 2013

Approval Signatures

Date

Date

OT January 2013

Date

OT January 2013

Date

OT January 2013

Date

OT January 2013

Date

OT January 2013

Date

# **TABLE OF CONTENTS**

| LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 4 |
|--------------------------------------------------------------------|----|
| 1. INTRODUCTION | 8 |
| 1.1 Study Design | 8 |
| 1.2 Study Objectives | 10 |
| 1.2.1 Primary Objective | 10 |
| 1.2.2 Resource Utilization and Patient Reported Outcome Objectives | 10 |
| 1.2.3 Exploratory Objective | 10 |
| 2. POPULATIONS FOR ANALYSIS | 10 |
| 2.1 Safety Population | 10 |
| 2.2 Efficacy Population. | 12 |
| 3. HYPOTHESES AND DECISION RULES | 13 |
| 4. INTERIM ANALYSIS | 13 |
| 4.1 Interim Analysis | 13 |
| 4.2 Data Safety Monitoring Board | 13 |
| 5. STUDY DEFINITIONS AND CONVENTIONS | |
| 5.1 Study Definitions | 13 |
| 5.2 Definition of Baseline Values | |
| 5.2.1 Change and Percent Change From Baseline | |
| 5.3 Visit Assignments | |
| 5.3.1 Study Start and End Dates | |
| 5.3.2 Visit Assignments for Efficacy Variables | 17 |
| 5.3.3 Visit Assignments for Safety Variables | |
| 5.3.4 Conventions for Missing Adverse Event Dates | |
| 5.3.5 Conventions for Missing Concomitant Medication Dates | 27 |
| 5.3.6 Conventions for Missing Previous Medication Dates | |
| 5.4 Calculation of Body Mass Index | 27 |
| 6. STATISTICAL METHODOLOGY | 28 |
| 6.1 Determination of Sample Size for the Long-term Safety Study | 28 |
| 6.2 Randomization and Stratification | |
| 6.3 Unblinding | 28 |
| 6.4 Methods for Handling Missing Data | 28 |
| 6.5 Patient Disposition | 28 |
| 6.6 Demographics and Baseline Disease Characteristics | |
| 6.6.1 Demographics | 29 |
| 6.7 Treatments and Medications | 31 |
| 6.7.1 Concomitant Medications and Procedures | 31 |
| 6.7.2 Study Drug Administration | 32 |
| 6.8 Safety Analyses | |
| 6.8.1 Safety Data Summary Grouping for Long-term Safety Study | |
| 6.8.2 Adverse Events | |
| 6.8.3 Laboratory Data | 41 |
| 6.8.4 ECG | 43 |

# Statistical Analysis Plan, Study C13008

| 6.8.5 Vital Signs | 44 |
|----------------------------------------------|----|
| 6.8.6 Immunogenicity Analysis | |
| 6.9 Exploratory Efficacy Analyses | |
| 6.9.1 General Methods | |
| 6.9.2 Exploratory Efficacy Endpoints | |
| 6.9.3 Exploratory Efficacy Analysis | |
| 6.10 Resource Utilization Outcomes | |
| 6.11 Patient-Reported Outcomes (PROs) | 48 |
| 7. CHANGES TO PLANNED ANALYSES FROM PROTOCOL | |
| 8. REFERENCES | 49 |

# Statistical Analysis Plan, Study C13008

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Term |
|--------------|-------------------------------------------|
| 5-ASAs | 5-aminosalicylates |
| AEs | adverse events |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| BUN | blood urea nitrogen |
| CD | Crohn's disease |
| CFR | Code of Federal Regulations |
| СНО | Chinese hamster ovary |
| $C_{min}$ | minimum plasma concentration |
| CMV | cytomegalovirus |
| CNS | central nervous system |
| CRP | C-reactive protein |
| CV | coefficient of variation |
| DSMB | data safety monitoring board |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| ELISA | enzyme-linked immunosorbent assay |
| EQ-5D | EuroQual |
| ET | early termination |
| GCP | good clinical practice |
| GI | gastrointestinal |
| h | hours |
| НАНА | human anti-human antibody |
| HBI | Harvey-Bradshaw Index |
| HCV | hepatitis C virus |
| HIV | human immunodeficiency virus |
| HLT | high level term |
| IAC | Independent Adjudication Committee |
| IB | Investigator's Brochure |
| IBD | inflammatory bowel disease |
| IBDQ | Inflammatory Bowel Disease Questionnaire |
| ICH | International Conference on Harmonisation |
| IEC | independent ethics committee |
| IFN | interferon |
| IL | interleukin |
| IRB | institutional review board |
| IV | intravenous |
| JCV | JC virus, a neurotropic DNA polyomavirus |
| IVRS | interactive voice response system |

# Statistical Analysis Plan, Study C13008

| Abbreviation | Term |
|--------------|----------------------------------------------------|
| MAdCAM-1 | mucosal addressin cell adhesion molecule-1 |
| MCS | mental component score |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Millennium | Millennium Pharmaceuticals, Inc. or its affiliates |
| MLN0002 | Vedolizumab |
| NSAID | nonsteroidal anti-inflammatory drug |
| PCS | physical component score |
| PD | pharmacodynamics |
| PK | pharmacokinetics |
| PML | progressive multifocal leukoencephalopathy |
| PT | Preferred Term |
| PVC | polyvinylchloride |
| QOL | quality of life |
| RAMP | Risk Assessment and Minimization for PML |
| RBC | red blood cell(s) |
| SAEs | serious adverse events |
| SF-36 | Short-Form 36 |
| SOC | System Organ Class |
| TB | tuberculosis |
| TNFα | tumor necrosis factor alpha |
| UC | ulcerative colitis |
| UCCS | Ulcerative Colitis Clinical Score |
| ULN | upper limit of normal |
| US | United States |
| VAS | visual analogue scale |
| WBC | white blood cell(s) |

Rationale for SAP amendment 2

The protocol was changed to include up to 400 additional patients with either ulcerative colitis or Crohn's disease who had not been previously treated with vedolizumab ("de novo patients"). The additional patients will increase the number of patients with exposure to vedolizumab and supplement the safety database to detect adverse events resulting from long-term vedolizumab administration that may not be detected in the year-long induction and maintenance studies. The addition of 400 patients allows for the detection of adverse events that occur at a prevalence of 0.1% to be detected with more than 85% likelihood, and events that occur at a prevalence of 1% to be detected with 99.99% likelihood. Importantly, the inclusion and exclusion criteria for the de novo patients are nearly identical to the criteria for patients who enrolled in Studies C13006, C13007, and C13011; study treatment and assessments are the same for these de novo patients as for rollover patients (those patients who enrolled in C13008 following participation in C13004, C13006, C13007, or C13011). The additional patients are enrolled at a subset of existing sites in select countries, including the United States (US).

In addition, with this protocol amendment, both rollover and de novo patients participating in C13008 will have access to vedolizumab until March 2016, or until vedolizumab is available in the country in which the patient resides, or until patient withdrawal, whichever comes first (unless the study is terminated early by the sponsor, as described in Section 11.12 of study protocol).

Another change to the protocol includes removal of JC virus DNA testing. When the vedolizumab pivotal studies were planned in 2008, it was unclear if JC virus DNA testing in the blood might be predictive of progressive multifocal leukoencephalopathy (PML) risk. More recently, controlled studies of natalizumab (which has a proven risk of PML) have conclusively demonstrated that detection of JC virus DNA in the blood is of no clinical utility in minimizing risk of PML. Therefore, monitoring for JC virus DNA in the blood has been discontinued.

Other changes to the protocol allow for the use of conventional, non-biological concomitant medications for IBD to be more consistent with standard clinical practice. Thus, patients are now allowed to start azathioprine, 6-mercaptopurine, methotrexate (methotrexate for CD only), or corticosteroids during the course of the study, even if they were not on these

### Statistical Analysis Plan, Study C13008

medications when enrolled in the study. In addition, oral corticosteroid regimens have been modified to be more consistent with individual patient needs, and the corticosteroid tapering requirement has been changed to a recommendation.

The definition of treatment failure that mandates withdrawal from the study has been modified to "long-term treatment failure" to more accurately reflect true treatment failure that occurs in clinical practice. Given the fluctuating natural history of inflammatory bowel disease (IBD), patients may be treated for short-term disease worsening with conventional therapies for IBD, as allowed per protocol, without being required to withdraw from the study. Accordingly, one of the criteria for the protocol-defined treatment failure, "disease worsening," that was based on disease activity indices (Harvey-Bradshaw Index and partial Mayo score), has been removed from the definition of long-term treatment failure. Importantly, patients are still required to be withdrawn if they require rescue medication or major surgery for the treatment of IBD.

### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) presents a detailed plan for the analyses of the long-term safety and efficacy study C13008. The analysis is designed to evaluate the safety profile of long-term vedolizumab treatment.

The objectives of this analysis are stated in Section 1.2, and a discussion of the analyses to be performed is provided in Section 6.8 through Section 6.11.

Reference materials for this SAP include Clinical Study Protocol C13008 (Amendment 10 of the protocol, dated 15 February 2012) and the accompanying data collection documents (Annotated Case Report Form [CRF], final version, dated 07 May 2012).

### 1.1 Study Design

This is an open-label, phase 3 study to support the long-term safety and efficacy of vedolizumab for the treatment of patients with moderate to severe ulcerative colitis (UC) or Crohn's disease (CD). All enrolled patients receive 300 mg vedolizumab administered every 4 weeks.

Most patients enrolling in this study have participated in a previous vedolizumab study (rollover patient).

- Patients with UC or CD who participated in the phase 2, open-label, long-term safety study (Study C13004), which includes up to 78 weeks of open-label treatment with vedolizumab.
- Patients who withdrew early from a phase 3 induction and maintenance study (Study C13006 [patients with UC] or Study C13007 [patients with CD]), which includes up to 50 weeks of blinded study treatment (vedolizumab or placebo). These patients must have withdrawn due to sustained non-response, disease worsening, or the need for rescue medications
- Patients who completed Study C13006 or Study C13007
- Patients who completed (through Week 10) Study C13011
- Waiver patient(s)

### Statistical Analysis Plan, Study C13008

For rollover patients, the first dose of vedolizumab in this study (Week 0) should occur no more than 9 weeks after the last dose of study drug in the previous study; the preferable period is within 3 to 5 weeks after the last dose in the previous study. Results of assessments from the last visit in the previous vedolizumab study are used to determine their eligibility to participate in this study. Baseline data are also obtained from the previous study, including medical history, disease history, demographics, tobacco use, and prior therapies.

In addition, up to 400 patients without previous treatment with vedolizumab are enrolled directly into this study (de novo patients). Patients with UC or CD must meet the inclusion/exclusion criteria for de novo patients (Section 5 of study protocol). Baseline data for these patients is obtained during the Screening period.

Following enrollment, all patients are administered 300 mg vedolizomab every 4 weeks for the duration of the study, followed by a 16-week post-treatment observation and safety assessment period. The total duration of MLN0002 treatment varies by patient based on continued benefit until March 2016, or until vedolizumab is available in the country in which the patient resides , or until patient withdrawal, whichever is sooner (unless the study is terminated early by the sponsor, as described in Section 11.12 of study protocol).

Patients may receive allowed concomitant medications for the treatment of IBD as detailed in Section 6.2.1 of study protocol, as determined by the principal investigator, at any time point during the study. Medications may be discontinued during the study, but if discontinuation is planned, it should be done prior to the first dose of vedolizumab.

It is strongly recommended that patients receiving oral corticosteroids begin an oral corticosteroid tapering regimen once they achieve clinical response or if, in the opinion of the investigator, they demonstrate sufficient improvement in clinical signs and symptoms.

Patients are withdrawn from the study for long-term treatment failure as described in the study definitions, or if they are not benefiting from therapy (see Section 6.2.3, Section 6.4.10, and Section 7.4 of study protocol).

All patients return 16 weeks after their last dose of MLN0002 for the Final Safety visit.

Safety assessments and efficacy assessments using the partial Mayo Score (for patients with UC) or the HBI score (for patients with CD) will be made throughout the treatment period.

# Statistical Analysis Plan, Study C13008

Detailed visit-by-visit study procedures and assessments are provided in the Schedule of Events and Section 7 of study protocol.

This trial is conducted in compliance with the protocol, good clinical practice (GCP), and the applicable regulatory requirements (including International Conference on Harmonisation [ICH] guidelines).

### 1.2 Study Objectives

### 1.2.1 Primary Objective

• To determine the safety profile of long-term vedolizumab treatment

### 1.2.2 Resource Utilization and Patient Reported Outcome Objectives

- To determine the effect of long-term vedolizumab treatment on time to major inflammatory bowel disease (IBD)-related events (hospitalizations, surgeries, and procedures)
- To examine the effect of long-term vedolizumab treatment on health-related quality of life (QOL) measurements

### 1.2.3 Exploratory Objective

• To obtain data regarding the effect of long-term vedolizumab treatment on maintaining clinical response and remission based on partial Mayo score (for patients with UC) and Harvey-Bradshaw Index (HBI) (for patients with CD)

### 2. POPULATIONS FOR ANALYSIS

There will be 2 analysis populations: the safety population and the efficacy population.

### 2.1 Safety Population

The safety population for this study is defined as all patients who receive any amount of

### Statistical Analysis Plan, Study C13008

vedolizumab in this study. Waiver patient(s) are excluded. The study safety population is used for all safety analyses.

Exposure for patients who first participated in Study C13004, C13006, C13007, or C13011 and who are now participating in the C13008 study, is evaluated from the first dose of vedolizumab in Studies C13004, C13006, C13007, and C13011.

For de novo patients, exposure is calculated from the first dose of vedolizumab in Study C13008.

Adverse events (AEs) are also evaluated from the first dose of vedolizumab in Studies C13004, C13006, C13007, and C13011 for the patients who received vedolizumab in Study C13004, C13006, C13007, or C13011. AEs are counted only during the time of vedolizumab administration, as follows:

- For patients who received placebo in Studies C13006, C13007, and C13011, AEs are counted from first dose of vedolizumab in the C13008 study.
- For patients who received vedolizumab in the induction phase and placebo in the maintenance phase, AEs are counted if the AE occurred between the first dose of vedolizumab and the last dose of vedolizumab in the induction phase.
- For patients who were in the placebo group in Study C13002, AEs are counted from the first dose of vedolizumab in the C13004 study.
- For patients who were in the vedolizumab group in Study C13002, AEs are counted from the first dose of vedolizumab in the C13002 study.
- For de novo patients, AEs are counted from the first dose of vedolizumab in the C13008 study.

Concomitant medications for patients who participated in Study C13004 and continue participating in Study C13008 are evaluated only for the C13008 experience, while the concomitant medications for patients who were in Studies C13006, C13007, and C13011 are evaluated following the administration of the first dose of vedolizumab in Studies C13006, C13007 and C13011.

### Statistical Analysis Plan, Study C13008

Concomitant medications for de novo patients are evaluated from first dose onwards of vedolizumab in C13008 Study.

Other safety data, such as laboratory parameters, vital signs, and electrocardiograms (ECGs), are evaluated only for the C13008 experience.

The safety data from patients who participate in Study C13008 as waiver patient(s) will be included in the listings but will not be represented in the summary tables and figures.

## 2.2 Efficacy Population

The efficacy population consists of all enrolled patients. However, to be included in an analysis at any specific time point, the patient must have had a post-baseline measurement for the time point. Additionally, to be included in a change from baseline analysis, the patient must have had a baseline measurement. Waiver patient(s) who receive any amount of vedolizumab in this study are excluded from the efficacy population.

The efficacy data for patients who were in Study C13006 or C13007 and continue participating in C13008 is analyzed from the first efficacy assessment in C13006 or C13007 for the maintenance intent-to-treat (ITT) population and non-ITT population. The maintenance ITT population has 3 treatment groups: placebo, vedolizumab every 4 weeks (Q4 wks) dosing, and vedolizumab every 8 weeks (Q8 wks) dosing. The non-ITT population has 2 treatment groups: placebo and vedolizumab every 4 weeks (Q4 wks).

The efficacy data for patients who were in Study C13011 and continue participating in Study C13008 is analyzed from the first efficacy assessment in C13011 by vedolizumab and placebo treatment groups.

The efficacy data for de novo patients is analyzed for the C13008 experience.

All efficacy analyses is performed for patients who completed the previous Study C13006 or C13007 (52 weeks completers) or C13011 (10 weeks completers) and those who terminated early (early termination) from C13006 and C13007.

The efficacy data for patients who participated in Study C13004 and continue participating in C13008 is not analyzed.

# Statistical Analysis Plan, Study C13008

The efficacy data from waiver patient(s) who participate in C13008 is included in the listings but is not included in the summary tables and figures.

The efficacy population is also used for all exploratory efficacy, resource utilization and patient reported outcome analyses.

### 3. HYPOTHESES AND DECISION RULES

The analyses are primarily descriptive in nature. Point estimations along with 95% confidence intervals are presented for important safety and efficacy parameters. No formal statistical hypothesis tests are performed.

### 4. INTERIM ANALYSIS

### 4.1 Interim Analysis

Two interim analyses will be conducted for safety at the time of BLA/MAA filing. Additional interim analyses on long-term safety data will be conducted for the Day 120 safety update(s).

### 4.2 Data Safety Monitoring Board

An independent data safety monitoring board (DSMB) reviews safety data from this study including, but not limited to, incidence of AEs and AEs of special interest (eg, infusion-related reactions, infections) on a regular basis and makes appropriate recommendations to Millennium. A statistical reporting organization has been designated by Millennium to provide the DSMB with essential safety data during the study. The DSMB does not review the efficacy data. The DSMB responsibilities, authorities, and procedures are documented in a DSMB charter.

# 5. STUDY DEFINITIONS AND CONVENTIONS

### 5.1 Study Definitions

Study terms and definitions are provided below.

# Pertaining to Patients with UC

| Term | Definition |
|---|---|
| Clinical Remission | A partial Mayo score of $\leq 2$ with no individual subscore $> 1$ . |
| Clinical Response | A decrease in the partial Mayo Score of at least 2 points and $\geq 25\%$ from baseline, with an accompanying decrease in rectal bleeding subscore of $\geq 1$ point from baseline or absolute rectal bleeding subscore of $\leq 1$ point |
| Rescue<br>Medication(s) | Any new medication to treat a new or unresolved luminal manifestation of ulcerative colitis (UC), with the following exceptions: oral and topical (rectal) 5-aminosalicylate (ASA) treatment oral corticosteroids per the guidelines outlined in Section 6.2.3 topical (rectal) corticosteroid enemas/suppositories azathioprine or 6-mercaptopurine; stable doses are recommended antibiotics antidiarrheals for control of chronic diarrhea oral probiotics (eg, Culturelle, Saccharomyces boulardii) |
| Long-term<br>Treatment Failure | Need for rescue medications, or major surgical intervention for treatment of UC, or a study drug-related adverse event leading to discontinuation from the study |
| Pertaining to Patients | with CD |
| Term | Definition |
| Clinical Remission | A HBI score ≤ 4 points |
| Clinical Response | $A \ge 3$ -point decrease in HBI score from baseline |
| Rescue<br>Medication(s) | Any new medication to treat a new or unresolved luminal manifestation of Crohn's disease (CD), with the following exceptions: • oral and topical (rectal) 5-ASA treatment |

Term Definition

- oral corticosteroids per the guidelines outlined in Section
   6.2.3
- topical (rectal) corticosteroid enemas/suppositories
- azathioprine, 6-mercaptopurine, or methotrexate; stable doses are recommended
- antibiotics
- antidiarrheals for control of chronic diarrhea
- probiotics (eg, Culturelle, *S. boulardii*)

Long-term
Treatment Failure

Need for rescue medications, or major surgical intervention for treatment of CD, or a study drug-related adverse event leading to discontinuation from the study

### **5.2** Definition of Baseline Values

For partial Mayo score, HBI, and QOL variables, the baseline value is defined as the last assessments before the first dose of study drug administration from each previous study in Studies C13006, C13007, and C13011. For medical history, UC/CD disease history, tobacco use, and prior therapies, the baseline value is also obtained from the previous studies. For demographics, the baseline value is defined as the last assessment before the first induction dose in Study C13006, C13007, or C13011 (see Section 6.6). For the analyses of UC or CD, overall phase 3 clinical response, changes in partial Mayo score, and changes in HBI are based on the baseline calculated in Study C13006, C13007, or C13011.

For safety analyses, such as laboratory values, vital sign measurements, and ECGs, baseline is defined as the value collected at the last visit before the first dose of vedolizumab in Study C13008. For human anti-human antibody (HAHA) and C-reactive protein (CRP) data, baseline values are also obtained from the previous studies.

For de novo patients, the baseline value is defined as the last assessment before the first dose of vedolizumab in Study C13008.

### **5.2.1** Change and Percent Change From Baseline

Change from baseline to any treatment study Week t is defined as follows:

$$C_t = M_t - M_{Baseline}$$

where:

- $C_t$  is the change from baseline at Week t
- M<sub>t</sub> is the measurement at Week t
- *M* <sub>Baseline</sub> is the measurement at baseline

Percent change from baseline to any maintenance treatment study Week t is defined as follows:

$$P_t = 100 \times (M_t - M_{Baseline}) / M_{Baseline}$$

The "Week t" to which the measurement belongs is determined using the conventions described in Section 5.3.

### 5.3 Visit Assignments

# 5.3.1 Study Start and End Dates

Enrollment is defined as the time at which the patient is entered into the Interactive Voice Response System (IVRS) for this study. Long-term safety study (C13008) treatment begins on the date of the first dose of study drug as recorded on the CRF.

Following enrollment, all patients are administered 300 mg vedolizumab every 4 weeks for the duration of the study, followed by a 16-week, post-treatment observation and safety assessment period. The total duration of vedolizumab treatment varies by patient based on continued benefit until March 2016, or until vedolizumab is available in the country in which the patient resides, or until patient withdrawal, whichever is sooner (unless the study is terminated early by the sponsor). The end of long-term treatment for patients who complete the study or who terminate early is defined as the date of the last known dose of vedolizumab during the C13008 study plus 16 weeks.

### **5.3.2** Visit Assignments for Efficacy Variables

<u>Week assignment</u>: Patients may not adhere strictly to the visit timing in the protocol. Therefore the designation of visits during the long-term safety is based on the day of evaluation relative to the start of the study rather than the nominal visit recorded in the CRF. Accordingly, the study is divided into continuous, mutually exclusive, analysis windows (Table 5-1), for the following efficacy measurements.

For efficacy parameters (partial Mayo score and HBI), if a patient has more than 1 score within a window, the assessment closest to the target day is used. In case of ties between observations located on different sides of the target day, the later assessment is used. If more than 1 score is available on the same day, the mean of the values is used.

Table 5-1 Day Windows: Partial Mayo Score and HBI Score for the Patients Who Were in Studies C13006 and C13007, and C13008 de novo patients

| Visit in C13006/7 | Target Day | Day Range |
|-------------------|------------|-----------|
| Week 2 | 15 | 2 - 21 |
| Week 4 | 29 | 22 - 35 |
| Week 6 | 43 | 36 - 56 |
| Week 10 | 71 | 57 – 84 |
| Week 14 | 99 | 85 - 112 |
| Week 18 | 127 | 113 - 140 |
| Week 22 | 155 | 141 - 168 |
| Week 26 | 183 | 169 – 196 |
| Week 30 | 211 | 197 – 224 |
| Week 34 | 239 | 225 - 252 |
| Week 38 | 267 | 253 - 280 |
| Week 42 | 295 | 281 - 308 |
| Week 46 | 323 | 309 - 336 |
| Week 50 | 351 | 337 - 357 |
| Week 52 | 365 | 358 - 392 |
| Visit in C13008 | Target Day | Day Range |
| Screening* | | |
| Week 0* | 1 | -14 |
| Week 4 | 29 | 15-42 |
| Week 8 | 57 | 43-70 |
| Week 12 | 85 | 71 – 112 |
| Week 20 | 141 | 113 – 168 |
| Week 28 | 197 | 169 – 224 |

Table 5-1 Day Windows: Partial Mayo Score and HBI Score for the Patients Who Were in Studies C13006 and C13007, and C13008 de novo patients

| | | - |
|----------|------|-------------|
| Week 36 | 253 | 225 – 280 |
| Week 44 | 309 | 281 - 336 |
| Week 52 | 365 | 337 - 392 |
| Week 60 | 421 | 393 – 448 |
| Week 68 | 477 | 449 – 504 |
| Week 76 | 533 | 505 - 560 |
| Week 84 | 589 | 561 – 616 |
| Week 92 | 645 | 617 - 672 |
| Week 100 | 701 | 673 - 728 |
| Week 108 | 757 | 729-784 |
| Week 116 | 813 | 785-840 |
| Week 124 | 869 | 841 - 896 |
| Week 132 | 925 | 897 – 952 |
| Week 140 | 981 | 953 - 1008 |
| Week 148 | 1037 | 1009 - 1064 |
| Week 156 | 1093 | 1065 - 1120 |
| Week 164 | 1149 | 1121 – 1176 |
| Week 172 | 1205 | 1177 – 1232 |
| Week 180 | 1261 | 1233 – 1288 |
| Week 188 | 1317 | 1289 – 1344 |
| Week 196 | 1373 | 1345 - 1400 |
| Week 204 | 1429 | 1401-1456 |
| Week 212 | 1485 | 1457-1512 |
| Week 220 | 1541 | 1513-1568 |
| Week 228 | 1597 | 1569-1624 |
| Week 236 | 1653 | 1625-1680 |
| Week 244 | 1709 | 1681-1722 |
| Week 248 | 1737 | 1723-1764 |
| Week 256 | 1793 | 1765-1820 |
| Week 264 | 1849 | 1821-1876 |
| Week 272 | 1905 | 1877-1932 |
| Week 280 | 1961 | 1933-1988 |
| Week 288 | 2017 | 1989-2044 |
| Week 296 | 2073 | 2045-2086 |
| Week 300 | 2101 | |
| | | 2087-2128 |
| Week 308 | 2157 | 2129-2184 |

Table 5-1 Day Windows: Partial Mayo Score and HBI Score for the Patients Who Were in Studies C13006 and C13007, and C13008 de novo patients

| Week 316 | 2213 | 2185-2240 |
|----------|------|-----------|
| Week 324 | 2269 | 2241-2296 |
| Week 332 | 2325 | 2297-2352 |
| Week 340 | 2381 | 2353-2408 |
| Week 348 | 2437 | 2409-2450 |
| Week 352 | 2465 | 2451-2492 |

<sup>•</sup> For de novo patients, screening and week 0 are from nominal visit.

Table 5-2 Day Windows: HBI Score for the Patients Who Were in Study C13011

| Visit in C13011 | Target Day | Day Range |
|-----------------|------------|-------------|
| Week 2 | 15 | 2 - 28 |
| Week 6 | 43 | 29-56 |
| Week 10 | 71 | 57-84 |
| Visit in C13008 | Target Day | Day Range |
| Screening* | | |
| Week 0* | 1 | -14 |
| Week 4 | 29 | 15-42 |
| Week 8 | 57 | 43-70 |
| Week 12 | 85 | 71 – 112 |
| Week 20 | 141 | 113 – 168 |
| Week 28 | 197 | 169 - 224 |
| Week 36 | 253 | 225 - 280 |
| Week 44 | 309 | 281 - 336 |
| Week 52 | 365 | 337 - 392 |
| Week 60 | 421 | 393 – 448 |
| Week 68 | 477 | 449 - 504 |
| Week 76 | 533 | 505 - 560 |
| Week 84 | 589 | 561 – 616 |
| Week 92 | 645 | 617 - 672 |
| Week 100 | 701 | 673 - 728 |
| Week 108 | 757 | 729-784 |
| Week 116 | 813 | 785-840 |
| Week 124 | 869 | 841 - 896 |
| Week 132 | 925 | 897 – 952 |
| Week 140 | 981 | 953 – 1008 |
| Week 148 | 1037 | 1009 - 1064 |

Table 5-2 Day Windows: HBI Score for the Patients Who Were in Study C13011

| Week 156 | 1093 | 1065 – 1120 |
|----------|------|-------------|
| Week 164 | 1149 | 1121 – 1176 |
| Week 172 | 1205 | 1177 – 1232 |
| Week 180 | 1261 | 1233 – 1288 |
| Week 188 | 1317 | 1289 – 1344 |
| Week 196 | 1373 | 1345 - 1400 |
| Week 204 | 1429 | 1401-1456 |
| Week 212 | 1485 | 1457-1512 |
| Week 220 | 1541 | 1513-1568 |
| Week 228 | 1597 | 1569-1624 |
| Week 236 | 1653 | 1625-1680 |
| Week 244 | 1709 | 1681-1722 |
| Week 248 | 1737 | 1723-1764 |
| Week 256 | 1793 | 1765-1820 |
| Week 264 | 1849 | 1821-1876 |
| Week 272 | 1905 | 1877-1932 |
| Week 280 | 1961 | 1933-1988 |
| Week 288 | 2017 | 1989-2044 |
| Week 296 | 2073 | 2045-2086 |
| Week 300 | 2101 | 2087-2128 |
| Week 308 | 2157 | 2129-2184 |
| Week 316 | 2213 | 2185-2240 |
| Week 324 | 2269 | 2241-2296 |
| Week 332 | 2325 | 2297-2352 |
| Week 340 | 2381 | 2353-2408 |
| Week 348 | 2437 | 2409-2450 |
| Week 352 | 2465 | 2451-2492 |

<sup>\*</sup> For de novo patients, screening and week 0 are from nominal visit.

# **5.3.3Visit Assignments for Safety Variables**

Table 5-3 Day Windows: JCV, Clinical Chemistry, and Hematology\*

| Visit in C13008 | Target Day | Day Range |
|-----------------|------------|-----------|
| Screening** | | |
| Week 4 | 29 | 2 - 56 |
| Week 12 | 85 | 57 – 112 |

Table 5-3 Day Windows: JCV, Clinical Chemistry, and Hematology\*

| Visit in C13008 | Target Day | Day Range |
|-----------------------|------------|----------------------------------|
| Week 20 | 141 | 113 – 168 |
| Week 28 | 197 | 169 – 224 |
| Week 36 <sup>a</sup> | 253 | 225 - 280 |
| Week 44 | 309 | 281 – 336 |
| Week 52 <sup>b</sup> | 365 | 337 - 392 |
| Week 60 | 421 | 393 – 448 |
| Week 68 <sup>a</sup> | 477 | 449 – 504 |
| Week 76 | 533 | 505 – 560 |
| Week 84 | 589 | 561 – 616 |
| Week 92 | 645 | 617 – 672 |
| Week 100 <sup>a</sup> | 701 | 673 – 728 (673 756) <sup>c</sup> |
| Week 108 | 757 | 729-784 |
| Week 116 | 813 | 785-840 (757-868) |
| Week 124 | 869 | 841 – 896 |
| Week 132 | 925 | 897 – 952 (869 – 980) |
| Week 140 | 981 | 953 – 1008 |
| Week 148 | 1037 | 1009 – 1064 (981- 1092) |
| Week 156 | 1093 | 1065 – 1120 |
| Week 164 | 1149 | 1121 – 1176 (1093 -1204) |
| Week 172 | 1205 | 1177 – 1232 |
| Week 180 | 1261 | 1233 – 1288 (1205 -1316) |
| Week 188 | 1317 | 1289 – 1344 |
| Week 196 | 1373 | 1345 – 1421 (1317 -1428) |
| Week 212 | 1485 | 1429-1540 |
| Week 228 | 1597 | 1541-1666 |
| Week 248 | 1737 | 1667-1792 |
| Week 264 | 1849 | 1793-1904 |
| Week 280 | 1961 | 1905-2030 |
| Week 300 | 2101 | 2031-2156 |
| Week 316 | 2213 | 2157-2268 |
| Week 332 | 2325 | 2269-2394 |
| Week 352 | 2465 | 2395-2535 |

<sup>\*</sup> JCV assessment, clinical chemistry and hematology are not conducted at Day 0. For baseline, the last measurement from the previous study (eg, C13004, C13006, C13007, or C13011) is used.

<sup>\*\*</sup> For de novo patients, screening and week 0 are from nominal visit.

a Schedule for CRP follows Weeks 36, 68, 100, 132, 164, and 196 visits window above.

b Schedule for coagulation follows Week 52, 104, and 152 visit window above.

c Windows in the brackets are for clinical chemistry and hematology in Years 3 and 4 only. . JCV testing

Table 5-3 Day Windows: JCV, Clinical Chemistry, and Hematology\*

| Visit in C13008 | Target Day | Day Range |
|-----------------|------------|-----------|

was discontinued per protocol amendment 8. No JCV testing beyond Week 196.

<u>Duplicate laboratory assessments</u>: If the same parameter is reported more than once on the same date, the mean of that parameter is used in the analyses. If a patient has more than 1 measure within a visit but on different dates, the assessment closest to the target day is used. In case of ties between observations located on different sides of the target day, the later assessment is used. In case of ties located on the same side of the target day (ie, more than 1 value for the same day), the mean of the values is used. For HAHA and CRP, if a patient has more than 1 measurement within the same study day, the highest value is used.

For JCV, if a patient has more than 1 measurement within an analysis window, the positive assessment value is chosen over a negative JCV value regardless of the target date. If more than 2 negative JCVs are within the same window, the 1 closest to the target date is used. If more than 2 positive JCVs are within the same window, the 1 with the higher titer value is chosen over the 1 with lower titer value. For duplicate vital sign parameters, the same rule as above is followed.

Table 5-4 Study Visit Windows: Vital Signs

| Target Day | Day Range |
|---|---|
| 29 | 2 - 42 |
| 57 | 43 - 70 |
| 85 | 71 - 98 |
| 113 | 99 – 126 |
| 141 | 127 – 154 |
| 169 | 155 - 182 |
| 197 | 183 - 210 |
| 225 | 211 - 238 |
| 253 | 239 - 266 |
| 281 | 267 – 294 |
| 309 | 295 - 322 |
| 337 | 323 - 350 |
| 365 | 351 - 378 |
| 393 | 379 - 406 |
| | 29<br>57<br>85<br>113<br>141<br>169<br>197<br>225<br>253<br>281<br>309<br>337<br>365 |

Table 5-4 Study Visit Windows: Vital Signs

| Visit in C13008 | Target Day | Day Range |
|-----------------|------------|-------------|
| Week 60 | 421 | 407 – 434 |
| Week 64 | 449 | 435 - 462 |
| Week 68 | 477 | 463 - 490 |
| Week 72 | 505 | 491 - 518 |
| Week 76 | 533 | 519 – 546 |
| Week 80 | 561 | 547 – 574 |
| Week 84 | 589 | 575 - 602 |
| Week 88 | 617 | 603 - 630 |
| Week 92 | 645 | 631 - 658 |
| Week 96 | 673 | 659 - 686 |
| Week 100 | 701 | 687 – 714 |
| Week 104 | 729 | 715 - 742 |
| Week 108 | 757 | 743 - 770 |
| Week 112 | 785 | 771 – 798 |
| Week 116 | 813 | 799 – 826 |
| Week 120 | 841 | 827 - 854 |
| Week 124 | 869 | 855 - 882 |
| Week 128 | 897 | 883 - 910 |
| Week 132 | 925 | 911 – 938 |
| Week 136 | 953 | 939 – 966 |
| Week 140 | 981 | 967 – 994 |
| Week 144 | 1009 | 995 - 1022 |
| Week 148 | 1037 | 1023 - 1050 |
| Week 152 | 1065 | 1051 - 1078 |
| Week 156 | 1093 | 1079 – 1106 |
| Week 160 | 1121 | 1107 - 1134 |
| Week 164 | 1149 | 1135 – 1162 |
| Week 168 | 1177 | 1163 – 1190 |
| Week 172 | 1205 | 1191 – 1218 |
| Week 176 | 1233 | 1219 – 1246 |
| Week 180 | 1261 | 1247 – 1274 |
| Week 184 | 1289 | 1275 – 1302 |
| Week 188 | 1317 | 1303 – 1330 |
| Week 192 | 1345 | 1331 - 1358 |
| Week 196 | 1373 | 1359 – 1386 |
| Week 200 | 1401 | 1387-1414 |
| Week 204 | 1429 | 1415-1442 |

Table 5-4 Study Visit Windows: Vital Signs

| Visit in C13008 | Target Day | Day Range |
|-----------------|------------|-----------|
| Week 208 | 1457 | 1443-1470 |
| Week 212 | 1485 | 1471-1498 |
| Week 216 | 1513 | 1499-1526 |
| Week 220 | 1541 | 1527-1554 |
| Week 224 | 1569 | 1555-1582 |
| Week 228 | 1597 | 1583-1610 |
| Week 232 | 1625 | 1611-1638 |
| Week 236 | 1653 | 1639-1666 |
| Week 240 | 1681 | 1667-1694 |
| Week 244 | 1709 | 1695-1722 |
| Week 248 | 1737 | 1723-1750 |
| Week 252 | 1765 | 1751-1778 |
| Week 256 | 1793 | 1779-1806 |
| Week 260 | 1821 | 1807-1834 |
| Week 264 | 1849 | 1835-1862 |
| Week 268 | 1877 | 1863-1890 |
| Week 272 | 1905 | 1891-1918 |
| Week 276 | 1933 | 19191946 |
| Week 280 | 1961 | 1947-1974 |
| Week 284 | 1989 | 1975-2002 |
| Week 288 | 2017 | 2003-2030 |
| Week 292 | 2045 | 2031-2058 |
| Week 296 | 2073 | 2059-2086 |
| Week 300 | 2101 | 2087-2114 |
| Week 304 | 2129 | 2115-2142 |
| Week 308 | 2157 | 2143-2170 |
| Week 312 | 2185 | 2171-2198 |
| Week 316 | 2213 | 2199-2226 |
| Week 320 | 2241 | 2227-2254 |
| Week 324 | 2269 | 2255-2282 |
| Week 328 | 2297 | 2283-2310 |
| Week 332 | 2325 | 2311-2338 |
| Week 336 | 2353 | 2339-2366 |
| Week 340 | 2381 | 2367-2394 |
| Week 344 | 2409 | 2395-2422 |
| Week 348 | 2437 | 2423-2450 |
| Week 352 | 2465 | 2451-2478 |

### Statistical Analysis Plan, Study C13008

\*For de novo patients, screening and week 0 are from nominal visit.

For parameters that are not listed in the above tables, data collected from scheduled visits are analyzed by the nominal visit week as labeled in the CRF. Data collected from unscheduled visits are presented in the listings, but not summarized in the pre-planned analysis. For example, IBDQ, SF-36, EQ-5D, and HAHA data are analyzed by the nominal visit week as labeled in the CRF.

<u>Duplicates in Quality of Life Parameters</u>: For handling partial and complete questionnaire data, when multiple records of the same type are present for a visit, the following conventions are used:

- If 1 complete score (all components and total [where applicable]) and 1 partial score (at least 1 missing component) are available for the same visit, the complete score is used—regardless of proximity to target date.
- If 2 partial scores are available, for overlapping components, the score from the date closest to the target date is given precedence for the given component. Components can be mixed from the 2 dates (if available components differ) and a new total calculated.
- If more than 1 complete score is available for the same visit, the data from the date closest to the target date is used.
- If partial scores are on separate dates but are the same proximity to the target date, the latest partial date is used.

### **5.3.4** Conventions for Missing Adverse Event Dates

Every effort is made to determine the actual onset date for the event or to obtain a reliable estimate for the onset date from the investigator.

For AEs or SAEs, a missing or incomplete onset date is imputed according to the following conventions:

1. If an onset date is missing, the derived onset date is calculated as the first non-missing valid date from the following list (in order of precedence):

### Statistical Analysis Plan, Study C13008

- First vedolizumab dose date
- Consent date (for SAEs only)
- 2. If an onset date is incomplete, the derived onset date is calculated by the following:
  - Missing day, but month and year present: the day is imputed as the 15<sup>th</sup> of the month. If the month and year are equal to the month and year of the first vedolizumab dose and the first vedolizumab dose occurs after the imputed date, the derived onset date is set equal to the first vedolizumab date. If the AE end date occurs before the imputed date, the derived onset date is set equal to the AE end date.
  - Missing day and month, but year present: the day and month is imputed as the 30<sup>th</sup> June of the year. If the year is equal to the year of the first vedolizumab dose and the first vedolizumab dose occurs after the imputed date, the derived onset date is set equal to the first vedolizumab date. If the AE end date occurs before the imputed date, the derived onset date is set equal to the AE end date.
  - If the imputed AE onset date occurs after the database lock date, the imputed AE onset date is imputed as the database lock date.

For AEs or SAEs, a missing or incomplete end date is imputed according to the following conventions:

- 1. If an end date is missing, the derived end date is imputed as the last assessment date, assuming that the last assessment occurs after the AE start. If the last assessment occurs before the AE start date, the derived end date is imputed as the AE start date.
- 2. If an end date is incomplete, the derived end date is calculated by the following:
  - Missing day, but month and year present: the day is imputed as the last date (for example February 2009 is imputed as 28 February 2009) of the month.
  - Missing day and month, but year present: the day and month is imputed as the 31<sup>st</sup> December of the year.
  - If the imputed AE end date occurs after the database lock date, the imputed AE end date is imputed as the database lock date.

### Statistical Analysis Plan, Study C13008

Missing dates for hospitalizations for UC or CD, colectomies (UC) or bowel surgeries (CD), and UC or CD procedures follow the same rules as previously defined.

### **5.3.5** Conventions for Missing Concomitant Medication Dates

Start and stop dates for all concomitant medications are collected on the CRF. However, in the case of missing or partial information in these dates, the following rules are used:

If the start date is missing or partial:

- If the day is missing, the start day is the first day of the month.
- If the month is missing, the start month is the month corresponding to 90 days before the first study medication date.
- If the year is missing, the start year is the year of the entry visit (or consent date, for those missing entry visit).
- If the entire date is missing, the start date is the date of first vedolizumab administration.

If the stop date is missing, partial, or "continuing:"

- If the day is missing, the stop day is the last day of the month reported.
- If the month is missing, the stop month is the month during which the last assessment occurred.
- If the year or the entire date is missing or if the medication is "continuing", the stop year is the year in which the last assessment occurred.

### **5.3.6** Conventions for Missing Previous Medication Dates

No dates are imputed for previous medications.

### 5.4 Calculation of Body Mass Index

Millennium calculates BMI as the ratio of patient's weight (in kilograms) to the square of the patient's height (in meters):  $BMI = kg/m^2$ .

### 6. STATISTICAL METHODOLOGY

# 6.1 Determination of Sample Size for the Long-term Safety Study

This is a phase 3 study to determine the long-term safety of vedolizumab (MLN0002) in patients with UC and CD. Most patients enrolled in this study have participated in a previous qualifying MLN0002 study as detailed in Section 4.1 (rollover patients). Up to 400 additional patients who have not been previously treated with vedolizumab may be enrolled (de novo patients) to supplement the safety database. The current estimate is that approximately 2200 patients in total will enter this study.

### 6.2 Randomization and Stratification

No randomization or stratification is planned for this study.

## 6.3 Unblinding

This is an open-label study; there is no blinding.

## 6.4 Methods for Handling Missing Data

All available safety and efficacy data are included in data listings and tabulations. No imputation of values for missing data are performed, except as described within this statistical analysis plan.

All patients who prematurely discontinue for any reason are considered censored for time to event type of analyses and endpoints.

### 6.5 Patient Disposition

Patient disposition is summarized by study:

- Patients who were in C13004 study,
- Patients who were in C13006 study,
- Patients who were in C13007 study
- Patients who were in C13011 study

### Statistical Analysis Plan, Study C13008

• De novo patients in C13008 study

In addition to the above 5 groups, safety data is also summarized by the following subgroups:

- By indication: UC and CD
- By prior TNF-α failures (Yes/No)

Data for waiver patients are not presented in the summary tables, but are displayed in the listings.

The disposition table displays the number of patients in:

- Safety Population
- Efficacy Population
- Prior TNF failure population
- Early termination from prior study
- Completed prior study
- Ongoing Patients
- Completed Long-term Safety Study
- Not Completing Long-term Safety Study, Primary Reasons

Patients who discontinued from the C13008 study are listed. This listing uses the safety population.

### 6.6 Demographics and Baseline Disease Characteristics

### 6.6.1 Demographics

For demographic characteristics, the baseline value is defined as the last assessment before the first induction dose of blinded study drug (C13006, C13007, or C13011) and the first dose of vedolizumab (C13004) or the assessment at screening for de novo patients.

### Statistical Analysis Plan, Study C13008

Demographic baseline data, such as age, gender, race, and ethnicity (Hispanic/Latino and non-Hispanic/Latino), body weight, BMI, and geographic region (as defined in Appendix 3) are summarized overall and by the 3 categories as defined in Section 6.5, using the safety population. Patient baseline age and BMI are summarized as continuous variables.

For baseline disease characteristics, UC- or CD-related medical and disease history and QOL baseline variables, the values are defined as the last assessments before the first dose of study drug administration in previous Studies C13004, C13006, C13007, and C13011. For de novo patients, the values at screening are used.

Disease-specific baseline disease characteristics are summarized by UC and CD indication, and by the categories as defined in Section 6.5.

Table 6-1 Summaries of UC/CD-Related Baseline Characteristics

| Characteristic | Summarized as | Categories |
|---|---|---|
| Duration of Crohn's Disease<br>(CD only) | Continuous | |
| Duration of Ulcerative Colitis (UC only) | Continuous | |
| Categorical Duration of<br>Ulcerative Colitis (UC only) | Categorical | < 1 year, ≥ 1- < 3 years, ≥3- < 7 years |
| Categorical Duration of Crohn's Disease ( CD only) | Categorical | < 1 year, $\geq$ 1- < 3 years, $\geq$ 3-7 years, missing |
| Patients with prior TNF $\alpha$ use | Categorical | Yes/No |
| Patients with prior TNF $\alpha$ failure | Categorical | Yes/No |
| Patients with TNF $\alpha$ and immunomodulator failure | Categorical | Yes/No |
| Patients with corticosteroid or immunomodulator | Categorical | Yes/No |
| Patients with only concomitant corticosteroid | Categorical | Yes/No |
| Patients with only concomitant immunomodulator | Categorical | Yes/No |
| Patients with concomitant corticosteroid and Immunomodulator | Categorical | Yes/No |
| Patients with concomitant corticosteroid | Categorical | Yes/No |
| Patients with concomitant immunomodulator | Categorical | Yes/No |
| HBI (CD only) | Continuous | |

Table 6-1 Summaries of UC/CD-Related Baseline Characteristics

| Characteristic | Summarized as | Categories |
|---|---|---|
| CRP (CD only) | Continuous | |
| Fistulizing Disease (CD only) | Categorical | Yes/No |
| Smoking Status | Categorical | Current Smoker |
| | | Nonsmoker |
| | | Former Smoker |
| Partial Mayo Score (UC only) | Continuous | |
| Baseline of Extraintestinal<br>Manifestations(UC only) | Categorical | Yes/No |
| Baseline of Extraintestinal<br>Manifestations(CD only) | Categorical | Yes/No |

For categorical characteristics, percent is calculated out of the total number of patients in the data set, overall and by subcohorts.

Duration of UC or CD is calculated as below:

(1 + C13008 first dose date – diagnosis date from C13004/006/007/011)/ 365.25.

For de novo patients, duration of UC or CD is calculated as (1 + C13008 first dose date – diagnosis date)/ 365.25.

Demographics are presented in listings for each patient in the safety population.

### 6.7 Treatments and Medications

#### 6.7.1 Concomitant Medications and Procedures

Concomitant medication is defined as medication, any amount of which is taken between the first and last day-(inclusive) of vedolizumab administration. Concomitant procedures are similarly defined.

Concomitant medications are summarized for the safety population by drug class (ATC Pharmacological subgroup), generic drug name, and patient categories as defined in Section 6.5. Concomitant medication use is also presented in listings.

Concomitant procedures are not coded, but presented in listings for each patient in the safety population.

### 6.7.2 Study Drug Administration

Patients receive open-label vedolizumab by intravenous (IV) infusion.

### 6.7.2.1 Extent of Exposure

Extent of exposure is defined as the number of complete infusions a patient receives. A patient must receive at least 75% of an infusion for it to be considered complete.

Exposure to study drug is defined as the number of days the patient received study drug based on the first and last doses regardless of in which study the beginning or end of dosing occurred. Given Q8 week dosing schedule, exposure also includes an additional 56 days after the last dose:

Exposure = (date of last infusion - date of first infusion) + 56

The cumulative distribution of the number of months on study drug (categorized by  $\geq 1$  month,  $\geq 6$  months,  $\geq 12$  months,  $\geq 18$  months,  $\geq 24$  months,  $\geq 30$  months, and  $\geq 36$  months) is provided as well as the cumulative distribution of the infusions.

The exposure presentations are provided for overall (CD and UC combined) and by indication. The overall vedolizumab experience includes the exposure to vedolizumab in all the trials (double-blind: C13006, C13007, and C13011 and open-label: C13002-C13004 and C13008).

The following rules are set up as referenced by the Request for Information FDA Advisory Committee April 2011.

#### General Rules:

- Last Dose Date in Induction is defined as the latest dose date entered into Inform, before the maintenance randomization date.
- Last Dose Date on Study is defined as the latest dose date entered into Inform.
- Methods are heavily reliant on data being entered into InForm.

### Statistical Analysis Plan, Study C13008

### Exposure Calculation Rules for Incorporating Up to 16 Week PK/PD Effect

### C13006/7 Patients

- Calculate exposure for C13006/7 and C13008 separately and sum.
- For C13006/7:
  - o If on placebo in Induction in C13006/7, then C13006/7 EXPOSURE = 0
  - o If on drug in Induction only (and not on drug in Maintenance):
    - Calculate C13006/7 End Exposure Date as min((Last Dose in Induction + 16 weeks), C13008 Start Date)
    - C13006/7 EXPOSURE = (C13006/7 End Exposure Date First Dose in Induction + 1)
  - o If on drug in Induction & Maintenance:
    - Calculate C13006/7 End Exposure Date as min (Last Dose in Maintenance + 16 weeks, C13008 Start Date)
    - C13006/7 EXPOSURE = (C13006/7 End Exposure Date First Dose in Induction + 1)
- For C13008:
  - End exposure date = min((Last Dose Date on C13008 + 16 weeks), Data Cutoff Date)
  - o C13008 EXPOSURE = (End Exposure Date-First Dose Date in C13008 + 1)
- TOTAL EXPOSURE = C13006/7 EXPOSURE + C13008 EXPOSURE

## C13011 Patients

- Calculate exposure for C13011 and C13008 separately and sum.
- For C13011:

### Statistical Analysis Plan, Study C13008

- o If placebo in C13011, then C13011 EXPOSURE = 0
- Calculate C13011 End Exposure Date as min ((Last Dose in Induction in C13011 + 16 weeks), C13008 Start Date)
- C13011 EXPOSURE = (C13011 End Exposure Date First Dose in Induction + 1)

### • For C13008:

- End exposure date = min((Last Dose Date on C13008 + 16 weeks), Data Cutoff Date)
- o C13008 EXPOSURE = (End Exposure Date-First Dose Date in C13008 + 1)
- TOTAL EXPOSURE = C13011 EXPOSURE + C13008 EXPOSURE

### C13002/4 Patients

For patients who have rolled over into C13008:

- For C13002/4:
  - Calculate C13002 End Exposure Date as min ((Last Dose in C13002 + 16 weeks), C13004 Start Date)
  - Calculate C13004 End Exposure Date as min ((Last Dose in C13004 + 16 weeks), C13008 Start Date)
  - If not in C13002 or on placebo in C13002, C13002/4 EXPOSURE = C13004
     End Exposure Date First Dose Date in C13004 + 1
  - If on drug in C13002, C13002/4 EXPOSURE = (C13004 End Exposure Date First Dose Date in C13004 + 1) + (C13002 End Exposure Date First Dose Date
    in C13002 + 1)
- For C13008:
  - Calculate C13008 End Exposure Date as min((Last Dose in C13008 + 16 weeks),
     C13008 Data Cutoff Date)

### Statistical Analysis Plan, Study C13008

C13008 EXPOSURE = (C13008 End Exposure Date-First Dose Date in C13008 + 1)

### TOTAL EXPOSURE = C13002/4 EXPOSURE + C13008 EXPOSURE

Exposure is also calculated incorporating up to 8 weeks (56 days). The same rules as above are applied but by adding 8 weeks instead of 16 weeks in the calculations.

# Exposure Calculation Rules Without Incorporating Up to 16 Week PK/PD Effect

In addition, exposure without incorporating up to 16 week PK/PD effect post last dose is calculated as below.

Use the exposure calculation rules above with the following modifications:

- 1. Do not add 16 weeks at any point in the calculations.
- 2. For patients C13006/7/11 on drug in induction only, calculate the end of exposure date as min (last dose date in induction + 4 weeks, C13008 start date).
- 3. For patients C13006/7 on drug in induction and maintenance, calculate the end of exposure date as min (last dose date in maintenance + 2 weeks, C13008 start date).

For de novo patients, the following rule is used to calculate exposure (in days):

- End exposure date = min((Last Dose Date on C13008 + 16 weeks), Data Cutoff Date)
- o C13008 EXPOSURE = (End Exposure Date-First Dose Date in C13008 + 1)

Extent of exposure for the long-term safety treatment is listed by patient.

### 6.8 Safety Analyses

Summaries of safety data such as Lab, JCV, RAMP, vital, PML checklist responses, and ECG are provided for data collected on patients during Study C13008 up to the final safety visit. These analyses are performed using the safety population.

Summary of AEs, SAE, and infections are based on the safety population as described in Section 2.1. In addition to incidence rates, rates of certain AEs, such as infections, are expressed in terms of time adjusted incidence rates (eg, events/person-year) to accommodate variable patient follow-up time and recurrent AEs within the same patient.
No statistical tests are performed.

#### 6.8.1 Safety Data Summary Grouping for Long-term Safety Study

AE incidence rates and other safety parameters are summarized for all C13002/4/6/7/8/11 patients, and by the patient groups defined in Section 6.5. In addition, incidence rates are summarized by CD and UC.

The comprehensive safety assessment as described in Section 8.7 of the C13008 Protocol Amendment 10 will be covered by the integrated safety summary that will have a separate analysis plan.

#### **6.8.2** Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA) is used for coding AEs. To summarize the number of patients with AEs, patients reporting the same event more than once has that event counted only once within each system organ class (SOC), high-level term (HLT), and preferred term (PT).

Key guidelines for the selection of AE incident rates for counting are as follows:

- 1. Where a patient has the same AE, based on preferred terminology, reported multiple times in a single analysis period, the patient is counted only once in the preferred terminology level in AE tables.
- 2. When a patient has the same AE, based on preferred terminology, reported multiple times in a single analysis phase, the following criteria, in order of precedence, are used to select the event to be included in summary tables.
  - Relationship to study medication
  - Intensity of event
  - Onset date and time (the earlier onset date and time are selected for the incident rates)
- 3. When reporting AE incident rates by intensity, the most intense event during the analysis phase is summarized, independent of relationship to study medication. For

#### Statistical Analysis Plan, Study C13008

these tables, the following criteria, in order of precedence, are used to select the event to be included in summary tables.

- Intensity of event
- Onset date and time (the earlier onset date and time are selected for the incident rates)

For any AE (serious or not), onset of the AE is determined using the Conventions outlined in Section 5.3.4.

In summaries by SOC, HLT, and PT, AEs are sorted by decreasing frequency of each PT, HLT, and SOC according to the incident rates. In summaries by PT, AEs are sorted by decreasing frequency within PT according to the incident rates.

#### **6.8.2.1** Treatment-Emergent Adverse Events

A treatment-emergent AE (TEAE) is defined as any new medical event/finding that occurs after the first vedolizumab administration in C13002/4/6/7/8/11 as recorded on the CRF.

#### **6.8.2.2** Time Adjusted Incidence Rates

To provide a benchmark for evaluation of AEs reported in the long-term safety study, a cohort study was performed on data from an external administrative database (HealthCore Integrated Research Database, HIRD<sup>TM</sup>), which includes a broad representation of patients on various therapies for IBD including biological agents. These analyses will provide estimates of the background rates of AEs of special interest.

For the analysis of the HIRD and Study C13008, the time adjusted incidence rate is defined as the number of patients experiencing an AE of interest divided by the person-time at risk. The amount of person-time will be truncated after a patient experiences an adverse event of special interest, although that patient will continue to contribute person-time for unrelated adverse events of special interest.

AE of special interest can be found in Appendix 8. The final list for AEs of special interest will depend on the results of Study C13008.

#### 6.8.2.3 All Adverse Events

AE incidence rates are summarized by SOC, HLT, PT, and by the groups defined in Section 6.5.

All reported AEs during the long-term safety study are listed by the groups defined in Section 6.5.

#### **6.8.2.4** Serious Adverse Events

Serious adverse event (SAE) incident rates are presented by SOC, HLT, PT, and by the groups defined in Section 6.5. In addition, related SAE incident rates are presented by SOC, HLT, PT, and by the groups defined in Section 6.5.

All SAEs are listed by the groups defined in Section 6.5.

#### **6.8.2.5** Deaths

All on-study deaths recorded on the AE page (outcome), or death page (with a death date and cause of death) of the CRF are considered in the analyses. All deaths are summarized by PT for the total patient group. All deaths are listed.

#### 6.8.2.6 Adverse Events Resulting in Discontinuation of Study Drug

AEs reported with an action taken of "discontinuation of study drug" are summarized by SOC, HLT, PT, and the groups defined in Section 6.5. Adverse events resulting in discontinuation of study are also summarized by SOC, HLT, PT, and CD/UC subgroups as defined in Section 6.5.

In addition, all AEs leading to discontinuation of study drug are listed.

#### **6.8.2.7** Adverse Events of Special Interest

Based on the mechanism of action of vedolizumab, certain adverse events and safety laboratories are of special interest. AEs of special interest include unusual or opportunistic infections, serious infections, and neoplasms. AEs of special interest are summarized by MedDRA SOC, HLT, and PT according to the groups defined in Section 6.5. Separately,

#### Statistical Analysis Plan, Study C13008

some AEs of special interest are also summarized by SOC, HLT, PT, and CD/UC subgroups as defined in Section 6.5.

The categories of adverse events of special interest and other planned analyses are as follows:

#### Infections

Summary tables of all serious infections and infections leading to discontinuation of study drug are presented. As vedolizumab is a local immunomodulator of the gastrointestinal tract, mucosal and gastrointestinal infections are also summarized separately. TEAE infections are also listed. Incidence of infections are summarized by the groups defined in Section 6.5. Infection rates are summarized by SOC, HLT, PT, and CD/UC subgroups as defined in Section 6.5.

Infections are also presented by time adjusted incidence rate (eg, events/person years).

Comparative rates of infection in patients who have not received concomitant immunomodulators or concomitant corticosteroids (monotherapy), patients who have received concomitant immunomodulators (eg, azathioprine, 6-mercaptopurine), and patients who have received concomitant corticosteroids (eg, prednisone, prednisolone), are reported.

#### Gastrointestinal Adverse Events

Subset analyses of all gastrointestinal AEs include all serious AEs and gastrointestinal AEs leading to discontinuations. Gastrointestinal AE incident rates are summarized by the patient groups defined in Section 6.5.

#### Infusion-Related Reactions/Immunogenicity

Infusion-related AEs are summarized by PT and the patient groups defined in Section 6.5. In addition, all AEs beginning on or 1 calendar day after the dates of study drug infusions are similarly analyzed. Comparative rates of infusion-related AEs are reported in HAHA-negative and HAHA-positive patients (see Section 6.8.6.3). Comparative rates of infusion-related AEs are also reported by CD/UC subgroups as defined in Section 6.5. Infusion-related AEs (investigator defined) are presented by preferred term.

#### Statistical Analysis Plan, Study C13008

Safety Related to Risk Management (RAMP Algorithm, JC Viremia, and Long-term Follow-up Data)

The protocol incorporates an active screening program to identify and manage any case of progressive multifocal leukencephalopathy (Protocol Section 10.5.3). This program is known as the Risk Assessment and Minimization for PML (or RAMP). In addition to the RAMP, plasma specimens were collected during the study and assayed for JC virus (JCV). However, JCV testing was discontinued per protocol amendment 8.

The results of the RAMP screening program are summarized for the patient groups defined in Section 6.5. Results of JCV testing are also summarized for the overall patient group. The RAMP algorithm findings are also listed.

Summary tables for long-term follow-up data are summarized.

Neoplasms (Benign, Malignant, and Unspecified)

All neoplasms are summarized overall, by patient groups, and by CD/UC subgroups as defined in Section 6.5.

#### **Liver Function Tests**

Descriptive statistics and shift tables for all liver function test results are reported, and all liver function abnormalities reported as AEs are summarized by the patient cohorts described in Section 6.5. In addition, the percentage of subjects who develop categorical increases ( $\leq 1$ , > 1 x ULN to  $\leq 2$  x ULN; > 2 x ULN to  $\leq 3$  X ULN, > 3 x ULN to  $\leq 5$  x ULN and > 5) in ALT, AST, or bilirubin are summarized. Individual narratives are written for patients with evidence of significant liver dysfunction.

#### Hematology

Descriptive statistics and shift tables for each subtype of white blood cell (ie, neutrophils, lymphocytes, monocytes, eosinophils, and basophils) are summarized by the patient groups defined in Section 6.5.

#### **6.8.2.8** Adverse Events in Special Groups

AEs by preferred term are presented separately based on the special groups listed below:

#### Statistical Analysis Plan, Study C13008

- Age ( $< 65, \ge 65 \text{ years}$ )
- Race (White, Black, Asian, and Other)
- Sex (Male, Female)
- Baseline disease activity (moderate [UC: Baseline Partial Mayo Score < 6, CD: CDAI < 330], severe [UC: Baseline Partial Mayo Score ≥ 6, CD: CDAI ≥ 330])</li>
- Body Weight (< 70 kg, 70-90 kg, > 90 kg)

#### 6.8.3 Laboratory Data

Unless otherwise specified, laboratory data obtained on and after Week 4 in the long-term safety study are included in the summary tables. Additionally, since laboratory tests will not be restricted to scheduled visits, Section 0 provides uniform visit windows to link each laboratory test to a scheduled visit. Assignment of patient treatment to a laboratory measurement is described in Section 0.

For the purposes of summarization in both the tables and listings, all laboratory values are converted to standardized units. If a lab value is reported using a non-numeric qualifier (eg, less than (<) a certain value, or greater than (>) a certain value), the given numeric value is used in the summary statistics, ignoring the non-numeric qualifier. All laboratory data are summarized by the patient groups defined in Section 6.5.

#### **6.8.3.1** Marked Laboratory Abnormalities

Laboratory abnormalities are evaluated based on marked abnormality (MA) criteria. Appendix 2 (Laboratory Abnormality Criteria) lists the predefined criteria for MAs. If both the baseline and on-treatment values of a parameter are beyond the same MA limit for that parameter, then the on-treatment value is considered an MA only if it is more extreme (farther from the limit) than the baseline value. If the baseline value is beyond the low MA limit and the on-treatment value is beyond the high MA limit (or vice versa), then the on-treatment value is considered a MA.

Laboratory MAs occurring during the long-term safety study are summarized. The directions of changes (high or low) in MAs are indicated in the tables. Additionally, for

#### Statistical Analysis Plan, Study C13008

each patient with an MA for a parameter, all the patient's values of that parameter over the long-term safety study are listed.

# 6.8.3.2 Changes from Baseline Values for Selected Laboratory Parameters over Time

The following hematology parameters and their changes from baseline values are summarized over all scheduled times of assessment, presenting n, means, medians, standard deviations and 95% CIs.

- hematocrit (changes from baseline)
- hemoglobin (changes from baseline)
- platelet count (changes from baseline)
- red blood cell (RBC) count (changes from baseline)
- white blood cell (WBC) count (changes from baseline)
- absolute neutrophil count (ANC) (changes from baseline)
- absolute lymphocyte count (changes and percent changes from baseline)
- absolute monocyte counts (changes and percent changes from baseline)
- absolute eosinophil counts (changes and percent changes from baseline)
- absolute basophil counts (changes and percent changes from baseline)

The following serum chemistry parameters and their change from baseline values are summarized over all scheduled times of assessment, presenting n, means, medians, standard deviations, and 95% CIs:

- total and direct bilirubin (changes from baseline)
- alanine aminotransferase (ALT) (changes from baseline)
- alkaline phosphatase (changes from baseline)

#### Statistical Analysis Plan, Study C13008

- aspartate aminotransferase (AST) (changes from baseline)
- amylase (changes from baseline)
- bicarbonate (changes from baseline)
- blood urea nitrogen (BUN) (changes from baseline).
- creatinine, serum (S<sub>cr</sub>) (changes from baseline)
- calcium (changes from baseline)
- glucose (changes from baseline)
- lipase (changes from baseline)
- magnesium (changes from baseline)
- phosphorus (changes from baseline)
- electrolytes sodium, potassium, chloride, (changes from baseline)
- total protein and albumin (changes from baseline)
- coagulation (changes from baseline)

Baseline is defined as the value collected at the last visit prior to the first dose of vedolizumab administration in C13008 study. The baseline and the visit window defined in Section 0 is followed for this calculation. For patients who were in C13004, the last measurement from C13004 is used for the baseline. For de novo patients, the assessments at screening are used for the baseline.

#### 6.8.4 ECG

Percent of subjects with abnormal ECGs are summarized by study visits. ECG abnormalities reported as AEs are summarized in the AE analysis as specified in Section 6.8.2.

#### 6.8.5 Vital Signs

The values and changes from baseline for heart rate, temperature, respiratory rate, and systolic and diastolic blood pressure are summarized by the patient groups defined in Section 6.5 at each scheduled time of assessment using the safety population. Vital sign abnormalities reported as AEs are summarized in the AE analysis as specified in Section 6.8.2.

#### 6.8.6 Immunogenicity Analysis

#### 6.8.6.1 Data Set Analyzed

HAHA baseline data is taken from the last measurements of the previous study (eg, C13004, C13006, C13007, or C13011) since HAHA is not measure on Day 0 of Study C13008. For de novo patients, the HAHA at screening is used for the baseline. Vedolizumab serum concentrations and HAHA data are summarized by study visits and by the patient groups defined in Section 6.5 using the safety population. Listings of vedolizumab and HAHA are also included. Serum concentration below limit of quantification is set to zero. No imputation is performed.

#### 6.8.6.2 HAHA Definitions

#### **Negative HAHA**

A sample that has been evaluated as negative in the HAHA screening assay is considered negative. Samples that are determined to be positive in the HAHA screening assay, but the result is not confirmed in the HAHA confirmatory assay is considered negative.

#### Positive HAHA

A sample that has been evaluated as positive in both the HAHA screening and confirmatory assays is considered positive.

#### Positive Neutralizing HAHA

A sample that has been evaluated as positive in the neutralizing HAHA assay is considered positive.

#### 6.8.6.3 Patient Status

**Baseline Positive** 

All patients who are HAHA positive from measurements from the previous study (eg, C13004, C13006, C13007, or C13011) are defined as baseline positive.

Patient HAHA status is further categorized and summarized as follows:

Negative

All patients who have no positive HAHA sample.

Positive

All patients who have at least 1 positive HAHA sample.

Persistent Positive

All patients who have 2 or more consecutive positive HAHA samples.

The maximum HAHA titer and percentage of subjects with each HAHA status are presented overall and by the patient groups defined in Section 6.5. Additional HAHA titer categories (eg, titer  $\geq 5, \geq 15, \geq 45, \geq 125, \geq 625$ , and  $\geq 3125$ ) are summarized if deemed appropriate.

#### 6.8.6.4 Effects of HAHA on Safety

Summary of overall AEs by HAHA status is presented. Summary of infusion-related AEs by HAHA status is also reported.

#### 6.9 Exploratory Efficacy Analyses

This section describes the analyses conducted on the exploratory efficacy, resource utilization, and patient-reported outcome endpoints.

#### 6.9.1 General Methods

The primary statistical focus for the exploratory efficacy analyses is on descriptive summary of efficacy endpoints rather than on formal analysis of the clinical data. Descriptive statistics, including 95% CIs, are provided for all clinical efficacy variables of interest.

#### Statistical Analysis Plan, Study C13008

The exploratory efficacy summaries are carried out using the baseline defined in Section 5.2. The exploratory efficacy analyses use the C13008 efficacy population.

#### 6.9.2 Exploratory Efficacy Endpoints

The following exploratory efficacy variables are summarized by study visits:

- HBI score (CD only)
- Proportions of HBI score  $\leq 4$ ,  $4 < \text{HBI score} \leq 7$  and HBI score  $\geq 7$
- Partial Mayo score (UC only)
- Proportions of Partial Mayo score  $\leq 2$ ,  $3 \leq$  partial Mayo score  $\leq 5$  and partial Mayo score  $\geq 6$
- CRP levels (CD only)

#### **6.9.3** Exploratory Efficacy Analysis

The descriptive statistics for observed values and change from baseline in CRP level, partial Mayo score (UC only) or HBI score (CD only), IBDQ score, SF-36 score, and EQ-5D score are summarized. The means of CRP level, partial Mayo score, and HBI score are plotted over time.

Table 6-2 describes the analyses for the exploratory efficacy objective.

Table 6-2 Summary of Analyses for Exploratory Objectives

| Variable | Subpopulation | Analysis Type |
|---|---|---|
| CRP level | CD | Tabulate descriptive statistics for observed values and change from baseline |
| Partial Mayo Score | UC | Tabulate descriptive statistics for observed values and change from baseline |
| Partial Mayo Score | UC | Proportions of Partial Mayo score $\leq 2$ , $3 \leq$ partial Mayo score $\leq 5$ and partial Mayo score $\geq 6$ over time |
| HBI Score | CD | Tabulate descriptive statistics for observed values and change from baseline |
| HBI Score | CD | Proportions of HBI score $\leq 4$ , $4 <$ HBI score $\leq 7$ and HBI score $> 7$ |

Table 6-2 Summary of Analyses for Exploratory Objectives

| Variable | Subpopulation | Analysis Type |
|---|---|---|
| CRP level | CD | Plot of mean observed values with 95% CI at each time point |
| Partial Mayo Score | UC | Plot of mean observed values with 95% CI at each time point |
| HBI Score | CD | Plot of mean observed values and with 95% CI at each time point |

Abbreviations: CD = Crohn's disease; CI = confidence interval; CRP = C-reactive protein; HBI = Harvey-Bradshaw Index; UC = ulcerative colitis.

A comprehensive efficacy assessment for long-term clinical response and clinical remission as measured by partial Mayo score for UC and by HBI for CD will be covered by the integrated summary of efficacy that will have a separate analysis plan.

#### 6.10 Resource Utilization Outcomes

Resources Utilization Outcomes collected in this study are as follows and are analyzed by CD or UC indication:

- Proportion of patients with CD-related hospitalization, bowel resection, or CD-related procedures(for CD patients)
- Proportion of patients with UC-related hospitalization, colectomies, or UC-related procedures (for UC patients)
- Time to CD-related hospitalization, bowel surgeries, or CD-related procedures (for CD patients)
- Proportion of patients with UC-related hospitalization, colectomies, or UC-related procedures (for CD patients)

For time-to-event analyses, Kaplan-Meier method is used for summarizing combined events.

Table 6-3 Summary of Analyses for Resource Utilization Objectives

| Variable | Population | Analysis Type |
|---|---|---|
| Time to combined CD-related events | Efficacy population CD patients | Kaplan Meier estimates along with 95% CI at 52, 100, 148,196 weeks and continued at weeks by approximately 1 year until the final safety visit |

Table 6-3 Summary of Analyses for Resource Utilization Objectives

| Variable | Population | Analysis Type |
|---|---|---|
| Time to combined UC-related events | Efficacy population UC patients | Kaplan Meier estimates-along with 95% CI at 52, 100, 148, 196 weeks and continued at weeks by approximately 1 year until the final safety visit |

Abbreviations: CD = Crohn's disease; CI = confidence interval; UC = ulcerative colitis.

#### 6.11 Patient-Reported Outcomes (PROs)

Patient-reported outcomes on quality of life collected in this study are as follows:

- Inflammatory Bowel Disease Questionnaire (IBDQ)
- Short Form-36 (SF-36)
- EuroQol (EQ-5D)

Patient-reported outcomes are analyzed using the efficacy population. The baseline value is the last measurement before the first dose of vedolizumab from the previous study (C13006, C13007 or C13011) as defined in Section 5.2.

Summary tables for patient-reported outcomes such as IBDQ include baseline and each scheduled visit for the endpoint under consideration.

Inflammatory Bowel Disease Questionnaire (IBDQ), SF-36, and EQ-5D are assessed at each scheduled visit. The mean changes from baseline in IBDQ total and subscale scores are presented along with 95% two-sided CIs for the differences in mean changes from baseline. In a similar manner, summaries of the changes from baseline in SF-36 summary scores physical component score (PCS) and mental component score (MCS), subscale scores, and EQ-5D utility and visual analogue scale (VAS) scores are provided.

Table 6-4 describes the tables and figures generated for the patient-reported outcomes objectives.

Table 6-4 Summary of Analyses for Patient-Reported Outcomes Objectives

| Variable | Imputation | Analysis Type |
|---|---|---|
| IBDQ (total) | Efficacy<br>Population | Changes from baseline at each scheduled visit, including mean and mean changes from baseline and 95% CI |
| IBDQ (subscales) | Efficacy<br>Population | Changes from baseline at each scheduled visits, including mean and mean changes from baseline and 95% CI |
| SF-36 (PCS and MCS) | Efficacy<br>Population | Changes from baseline at each scheduled visits, including mean and mean changes from baseline and 95% CI |
| SF-36 (subscales) | Efficacy<br>Population | Changes from baseline at each scheduled visits, including mean and mean changes from baseline and 95% CI |
| EQ-5D Utility | Efficacy<br>Population | Changes from baseline at each scheduled visits, including mean and mean changes from baseline and 95% CI |
| EQ-5D VAS | Efficacy<br>Population | Changes from baseline at each scheduled visits, including mean and mean changes from baseline and 95% CI |

#### 7. CHANGES TO PLANNED ANALYSES FROM PROTOCOL

Patients who previously participated in the phase 2, open-label, long-term safety study (Study C13004) are part of the integrated safety analysis for Study C13008. Exposure, AE, and concomitant medication data from all patients who previously participated in Study C13004 are analyzed in Study C13008.

#### 8. REFERENCES

- 1. Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. December, 2004
- 2. Lachin, J.M., Biostatistical Methods, The Assessment of Relative Risks, 2000, *Wiley Serious in Probability and Statistics*

### **APPENDICES**

### APPENDIX 1 TABLES AND FIGURES

Tables and Figures will be provided upon request.

#### APPENDIX 2 LABORATORY ABNORMALITY CRITERIA

Table A2.1 provides the criteria for assessing marked abnormalities in safety laboratory parameters with thresholds based on grade 2 moderate intensity levels from the Division of AIDS table for grading the severity of adult and pediatric adverse events (December, 2004). As stated in Section 6.11.2.1, if both the baseline and on-treatment values of a parameter are beyond the same MA limit for that parameter, then the on-treatment value is considered a MA only if it is more extreme (farther from the limit) than was the baseline value.

| Table A2.1: Marked Abnormality Criteria for Safety Laboratory Parameters | | | | |
|---|---|---|---|---|
| Parameter | Test Code | Units | Direction of Change | Marked Abnormalities |
| HEMATOLOGY | | | | |
| Hemoglobin | НВ | g/L | Low Only | $\leq 70~\mathrm{g/L}$ |
| Absolute Lymphocyte<br>Count | LYMPH | 10E9 | Low Only | <0.5 X10E9 |
| Leukocytes | WBC | 10E9 | Low Only | Absolute Value < 2.0X10E9 |
| Platelets | PLT | 10E9 | Low Only | <75.0X10E9 |
| Absolute Neutrophil Count | ANC | 10E9 | Low Only | <1.0X10E9 |
| Prothrombin Time | PT | % | High Only | >1.25 x ULN |
| CHEMISTRIES | | | | |
| SGPT | ALT | ULN | High Only | >3.0 x ULN |
| SGOT | AST | ULN | High Only | >3.0 x ULN |
| Bilirubin | BILI | ULN | High Only | >2.0 x ULN |
| Amylase | AMYL | ULN | High Only | >2.0 x ULN |
| Lipase | LIP | ULN | High Only | >2.0 x ULN |
| Serum Creatinine | CREAT | ULN | High Only | >2.0 x ULN |

### APPENDIX 3 GEOGRAPHIC REGIONS

| Region | | Countries | |
|--------------------------|-----------------|-------------|----------------|
| North America | Canada | Puerto Rico | United States |
| Western/ Northern Europe | Austria | Belgium | Denmark |
| | France | Germany | Iceland |
| | Ireland | Italy | Netherlands |
| | Norway | Portugal | Spain |
| | Sweden | Switzerland | United Kingdom |
| Central Europe | Czech Republic | Greece | Hungary |
| | Poland | Romania | Serbia |
| | Slovak Republic | | |
| Eastern Europe | Bulgaria | Estonia | Israel |
| | Latvia | Malta | Russia |
| | Turkey | Ukraine | |
| Africa/Asia / Australia | Australia | Hong Kong | India |
| | New Zealand | South Korea | Malaysia |
| | Taiwan | China | Singapore |
| | South Africa | | |

### APPENDIX 4 MAYO SCORE CALCULATION WORKSHEET

## Complete and Partial Mayo Scoring "Points to Remember"

The Mayo Score is widely used in clinical trials to assess Ulcerative Colitis disease activity. It is a combination of two patient-reported and two physician-determined components. The Partial Mayo Score includes only the Stool Frequency, Rectal Bleeding, and PGA subscores. (Does not include endoscopy)

#### **Sub Scores**

| Sub Scores | |
|---|---|
| Stool Frequency (Patient) | Stool frequency WILL: Be |
| 0 = Normal number of stools for this patient | derived from patient reported diary data in IVRS and will be the average of 3 days prior to visit |
| 1 = 1 to 2 stools more<br>than normal<br>2 = 3 to 4 stools more<br>than normal | ➤ Be variable from patient to patient. Instruct patients to set the baseline of "normal" to whatever is "normal" for them. (eg, A patient normally has 1 stool per day and today has had 4 stools. Therefore the patient has had 3 more than "normal", which yields a value of 2 for that day) |
| 3 = 5 or more stools more than normal | Be defined as the passage of solid or liquid fecal material. Episodes of incontinence count. A non-productive trip to the bathroom or the simple passage of gas DO NOT COUNT as a stool. |
| Rectal Bleeding | Rectal bleeding WILL: |
| (Patient) $0 = \text{No blood seen}$ | Be derived from patient reported diary data in IVRS and will be the average of 3 days prior to visit |
| 1 = Streaks of blood with<br>stool less than half the<br>time | Represent the most severe bleeding of the day. Hemorrhoidal bleeding DOES NOT COUNT. |
| 2 = Obvious blood with<br>stool most of the time<br>3 = Blood alone passes | |
| Findings on Endoscopy (Physician) 0 = Normal or inactive disease 1 = Mild disease (erythema, decreased vascular pattern, mild friability) 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions) 3 = Severe disease (spontaneous bleeding, ulceration) | Findings on Endoscopy WILL: Be documented by photographic evidence Be classified by the worst affected segment if mucosal appearance varies Be characterized as follows Moderate: Bleeds to touch (forceps applied to colonic mucosa for 1 second) Severe: Bleeds spontaneously Endoscopy should be performed by the same endoscopist for any given patient |
| Physician's Global Assessment (Physician) 0 = Normal | Physician's Global Assessment WILL: > Be based on the patient's overall status on the day of visit > Reflect how the patient is doing at present. Assessment SHOULD NOT reflect past disease severity or complexity or the number/kinds of medications the patient is |

#### Statistical Analysis Plan, Study C13008

| 1 = Mild disease | | receiving. |
|---|---|---|
| 2 = Moderate disease | > | Be based on the |
| 3 = Severe disease | | • Other 3 components of the Mayo score |
| | | • Patient's recollection of abdominal discomfort and general sense of well-being |
| | | • Patient's performance status, fecal incontinence, and mood |
| | | <ul> <li>Physician's observations and physical exam findings</li> </ul> |
| | > | Reflect disease activity, NOT disease severity (eg. Do not automatically give a high PGA to patients with pancolitis or severe/complicated disease, or patients requiring multiple medications.) |

- If calculated manually, subscores should be rounded to the nearest integer.
- The Mayo score is equal to the sum of the subscores.

### APPENDIX 5 AES OF SPECIAL INTEREST

- Gastrointestinal Events
  - Use SOC of GASTROINTESTINAL DISORDERS to flag
- Malignancies
  - Use SOC of NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) to flag
- Infections
  - Use SOC of INFECTIONS AND INFESTATIONS to flag
- Infusion Related Reactions
  - Analysis for these AEs will occur on two levels:
    - Investigator defined Infusion Related Reactions (as indicated on the AE CRF)
    - All AEs that occur on or one calendar day after the infusion date.

### APPENDIX 6 PRIOR THERAPIES

| | Systemic<br>Corticosteroids | Immunomodulators | Anti TNF |
|---|---|---|---|
| CRF Label | Systemic<br>Corticosteroids | Azathioprine/ 6-Mercaptopurine | Infliximab |
| | | Methotrexate | Adalimumab |
| | | | Certolizumab |

### APPENDIX 7 PATIENT REPORTED OUTCOMES

| Table A7.1: | Patient Reported Outcomes – IB | DQ, SF-36 and EQ-5D |
|---|---|---|
| Variable | | |
| SF-36 | Sub-score | Calculation |
| | Physical Functioning (raw score) | Sum of (Q3a, Q3b,Q3c,Q3d,Q3e,Q3f,Q3g,Q3h,Q3i, Q3J) |
| | Role Physical (raw score) | Sum of (Q4a, Q4b, Q4c, Q4d) |
| | Bodily Pain (raw score) | Sum of (Q7,Q8) |
| | General Health (raw score) | Sum of (Q1, Q11a, Q11b, Q11c, Q11d) |
| | Vitality (raw score) | Sum of (Q9a, Q9e, Q9g, Q9i) |
| | Social Functioning (raw score) | Sum of (Q6, Q10) |
| | Role-Emotional (raw score) | Sum of (Q5a, Q5b, Q5c) |
| | Mental Health (raw score) | Sum of (Q9b,Q9c,Q9d,Q9f,Q9h) |
| Note | missing at a visit, the MEA imputed as the value for the | above, if 50% or less of the component score is N of the remaining component score will be emissing component score. If more than 50% of sing for the item, the imputed value will be set to |
| | Physical Functioning (S-score) | (PF score -10)/20*100 |
| | Role Physical (S- score) | (RP score -4)/16*100 |
| | Bodily Pain (S- score) | (BP score-2)/10*100 |
| | General Health (S- score) | (GH score -5)/20*100 |
| | Vitality (S- score) | (VT score -4)/16*100 |
| | Social Functioning (S-score) | (SF score -2)/8*100 |
| | Role-Emotional (S- score) | (RE score -3)/12*100 |
| | Mental Health (S- score) | (MH score -5)/20*100 |
| | Physical Functioning (Z-score*) | (PF - 83.29094)/23.75883 |
| | Role Physical (Z-score) | (RP-82.50964)/25.52028 |
| | Bodily Pain (Z-score) | (BP-71.32527)/23.66224 |
| | General Health (Z-score) | (GH-70.84570)/20.97821 |
| | Vitality (Z-score) | (VT-58.31411)/20.01923 |
| | Social Functioning (Z-score) | (SF-84.30250)/22.91921 |
| | Role-Emotional (Z-score) | (RE-87.39733)/21.43778 |

| Table A7.1: | Patient Reported Outcomes – IB | DQ, SF-36 and EQ-5D |
|---|---|---|
| Variable | | |
| | Mental Health (Z-score) | (MH-74.98685)/17.75604 |
| | Aggregated physical score | $PHYS = (PF_Z*0.42402) + (RP_Z*0.35119) + (RP_Z*0.35119)$ |
| | Se semi F years | BP Z*0.31754)+(GH Z*0.24954)+( |
| | | VT_Z*0.02877) +( SF_Z*0.00753*(-1))+( |
| | | RE Z* 0.19206*(-1)) + (MH Z*0.22069*(-1)) |
| | Aggregated Mental score | MENT = (PF Z*0.22999*(-1)) + |
| | | (RP Z*0.12329* |
| | | (-1)) +( BP Z*0.09731*(- |
| | | 1))+(GH_Z*0.01571*(-1))+ (VT_Z*0.23534) +( |
| | | SF_Z*0.26876)+( RE_Z* 0.43407) + |
| | | (MH_Z*0.48581) |
| | If less than or equal to 4 Z- | scores are missing, the average of the remaining Z |
| Note | scores will be used to comp | oute the value for the missing component score. If |
| Note | more than 4 Z scores are m | issing, the aggregate mental or physical will be set |
| | to missing. | |
| IBDQ | Sub-score | Calculation |
| | IBDQ Bowel symptoms | Sum of (Q1, Q5, Q9, Q13, Q17, Q20, Q22, Q24, |
| | score | Q26, Q29), Ranging from 10 to 70, 10 questions |
| | IBDQ Emotional function | Sum of (Q3, Q7, Q11, Q15, Q19, Q21, Q23, |
| | score | Q25, Q27, Q30, Q31, Q32), Ranging from 12 to |
| | | 84, 12 questions |
| | IBDQ Social function | Sum of (Q4, Q8, Q12, Q16,Q28), Ranging from |
| | score | 5 to 35, 5 questions |
| | IBDQ Systemic symptoms | Sum of (Q2, Q6, Q10, Q14,Q18), Ranging from |
| | score | 5 to 35, 5 questions |
| | For each component score | above, if 50% or less of the component score is |
| | | N of the remaining component score will be |
| Note | - | e missing component score. If more than 50% of |
| | the component score is mis | sing for the item, the imputed value will be set to |
| | missing. | |
| | IBDQ score | Sum of (bowel, emotion, social, system) |
| Note | | ore is missing at a visit, the imputed value will be |
| | set to missing | |
| EQ-5D | Sub-score | Calculation |
| | EQ5D Mobility | Ranging from 1 to 3 |
| | component score | |
| | EQ5D self-care | Ranging from 1 to 3 |
| | component score | |
| | EQ5D usual activities | Ranging from 1 to 3 |
| | component score | |
| | EQ5D Pain/discomfort | Ranging from 1 to 3 |

| Table A7.1: Patient Reported Outcomes – IBDQ, SF-36 and EQ-5D | | |
|---|---|---|
| Variable | | |
| | component score | |
| | EQ5D anxiety/depression | Ranging from 1 to 3 |
| | component score | |
| Note | the remaining component so | If 2 or less out of 5 of the components are missing at a visit, the MEAN of the remaining component score will be imputed as the value for the missing component score. If 3 or more components are missing, the imputed value will be set to missing. |
| EQ5D VAS | , | On a scale of 0 to 100, where 0 is the worst imaginable health state and 100 is the best imaginable health state. |

<sup>\*</sup> Z-scores formula are described in the SC-36 Manual

### Statistical Analysis Plan, Study C13008

### APPENDIX 8 AES OF SPECIAL INTEREST

| Infections |
|--------------------------------------------------------------|
| Bacterial pneumonia |
| Bacteremia |
| Sepsis |
| Pneumocystis jiroveci (carinii) pneumonia |
| Pyelonephritis |
| Herpes zoster |
| Progressive multifocal leukoencephalopathy |
| Tuberculosis |
| Histoplasmosis |
| Listeria meningitis |
| Mycobacteria avium complex |
| Candidiasis |
| Herpes simplex |
| Dental abscesses/periodontitis |
| Rectal or peritoneal abscesses |
| Salmonella septicemia |
| Cryptosporidiosis |
| C. difficile diarrhea/colitis |
| CMV colitis |
| Urinary tract infection |
| Giardiasis |
| Cellulitis |
| Viral meningitis |
| Cancer |
| All primary solid tumors |
| Lymphatic and hematopoietic malignancies |
| Lymphosarcoma and reticulosarcoma |
| Marginal zone lymphoma |
| Hodgkin's disease |
| Other malignant neoplasms of lymphoid and histiocytic tissue |
| Peripheral t-cell lymphoma |
| Multiple myeloma and immunoproliferative neoplasms |
| Lymphoid leukemia |

Lymphoid leukemia

Myeloid leukemia

Monocytic leukemia

Other leukemia

Digestive tract

Oropharyngeal

| Statistical Analysis Plan, Study C13008 |
|---|
| Esophagus |
| Stomach |
| Small intestine |
| Colon |
| Rectum, anus |
| Intrahepatic bile ducts |
| Gall bladder |
| Pancreas |
| Retroperitoneum and peritoneum |
| Other |
| Cervical carcinoma |
| Melanoma |
| B-cell lymphoma |
| Cervical dysplasia |
| Gastrointestinal |
| Intestinal obstruction/stenosis |
| Abdominal abscesses |
| Abscess of anal and rectal regions |
| Campylobacter gastroenteritis |
| Salmonella gastroenteritis |
| Viral gastroenteritis |
| Intestinal/gastric perforation |
| Miscellaneous |
| Deep venous thrombophlebitis |
| Pulmonary embolus |
| Stroke |
| Congestive heart failure and/or Stevens-Johnson syndrome/toxic epidermal necrolysis |
| Erythema multiforme |
| Stevens-Johnson syndrome/Toxic epidermal necrolysis |
| Acute myocardial infarction |
| Kidney stones |
| Acute renal failure/renal insufficiency (excluding chronic) |

Angioedema